CLINICAL TRIAL: NCT03190525
Title: CLinical Decision-making, Prognosis, quAlity of Life and Satisfaction With caRe in patIents With Relapsed/refracTory Multiple mYeloma (CLARITY)
Brief Title: Clinical Decision-making, Prognosis, Quality of Life and Satisfaction in Relapsed/Refractory Multiple Myeloma
Acronym: CLARITY
Status: Active, not recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: QoL-MM1016
Record Dates: First submitted 2017-06-12; First posted 2017-06-16 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Multiple Myeloma patients
  Interventions: Other: Quality of life questionnaires

INTERVENTIONS:
Other: Quality of life questionnaires — QLQ-C30

SUMMARY:
The primary objective is overall survival (OS) as predicted by baseline self-reported EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30) fatigue scale ratings, independently from other prognostic factors for OS in multiple myeloma (MM), including the clinically-based prognostic frailty score.

DETAILED DESCRIPTION:
While quality of life (QoL) and other types of patient-reported Outcomes (PROs) can be crucial in the management of RRMM patients, a perusal of the literature indicates a dearth of information in this area. PRO is defined by the US Food and Drug Administration (FDA) as "a measurement based on a report that comes directly from the patient (i.e., study subject) about the status of a patient's health condition without amendment or interpretation of the patient's response by a clinician or anyone else. A PRO can be measured by self-report or by interview provided that the interviewer records only the patient's response. Until now the few studies that have included PRO data have been conducted in newly diagnosed MM patients enrolled in randomized controlled trials (RCTs).

For the purpose of this protocol, we have conducted a systematic review of PRO studies conducted in RRMM patients receiving treatments with either Imunomodulatory agents (IMiDs) or Proteasome inhibitors (PIs). The search was conducted for studies published from January, 1990 to July, 2015 and yielded only eight studies published within this timeframe. Three studies dealt with bortezomib based regimens, two with thalidomide, and the remaining studies with carfilzomib, pomalidomide, and lenalidomide. In all these studies PROs were considered as secondary outcomes and in four this was analyzed in the context of RCTs.

Despite enhanced disease control, none of the current novel agents, either IMiDs or PIs are free of significant toxicities, which frequently persist after completing treatment and continue to impair patient's daily functioning over the long-term period. Also, it is important to consider the poor prognosis for many of these patients. For example, patients who fail first-line PIs or IMiDs have been shown to report an average life expectancy of 9 months from the time of becoming refractory to PIs and IMiDs. Maintaining a "good" or "acceptable" level of QoL and lowering symptom burden over the longest possible period of time is a main goal of treatment for RRMM patients. Therefore, considering the paucity of QoL evidence-base data, CLARITY is designed to expand on some key understudied areas in this population that are broadly summarized in the next two paragraphs.

ELIGIBILITY:
Inclusion Criteria:

* MM patients who have received at least 1 prior line of therapy and are considered as RRMM according to IMWG criteria.
* Adult patients (≥ 18 years old).
* Written informed consent provided.
* Patients who have been enrolled onto other study therapy protocols are also eligible.
* Having a full baseline PRO evaluation completed.
* All data a available to calculate the frailty score.

Exclusion Criteria:

* Having any kind of psychiatric disorder or major cognitive dysfunction hampering the provision of informed consent.
* Having reported any grade ≥3 adverse event within two weeks prior to study entry.
* Having received more than 5 lines of therapies.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Considering the observational nature of study and fact that we aim to provide data on RRMM patients from the real-world setting, we have set up very broad inclusion criteria. Patients enrolled in clinical trials are still eligible for this protocol. Possible participation in a clinical trial at the time of entry in this study will be recorded and used for sensitivity analysis.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2017-11-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective is overall survival (OS) as predicted by baseline self-reported EORTC QLQ-C30 fatigue scale ratings, independently from other prognostic factors for OS in MM, including the clinically-based prognostic frailty score. | 30 months from study entry

SECONDARY OUTCOMES:
To devise a patient-centered frailty score for RRMM patients. | 30 months from study entry
To investigate the prognostic value of the frailty score in the setting of RRMM. | 30 months from study entry
To investigate QoL over time (outcome measures: EORTC QLQ-C30 and QLQ-MY20) by type of treatment and examine factors that contribute the most in maintaining baseline QoL levels. | 30 months from study entry
To investigate relationship between satisfaction with information provision (outcome measure: EORTC INFO-25) and QoL outcomes (outcome measures: EORTC QLQ-C30 and QLQ-MY20). | 30 months from study entry
To assess patients' preferences for involvement in treatment decision-making and the relationships between preferences and patient characteristics. | 30 months from study entry
To assess and compare the baseline self-reported EORTC QLQ-C30 fatigue scale ratings, between those RRMM patients who had received only one line of treatment (1 line) versus more than one line of treatment (>1 line) at study entry | 30 months from study entry

CONTACTS AND LOCATIONS:
Overall Officials: Maria Teresa Petrucci, MD, Principal Investigator — Roma Sapienza; Fabio Efficace, Study Chair — GIMEMA Foundation
Locations (35):
- Italy (34):
  - Azienda Ospedaliero - Universitaria Ospedali Riuniti Umberto I - G.M. LANCISI - G. SALESI, Ancona
  - S. Orsola Malpighi, Bologna
  - Divisione di Ematologia Ospedale A. Perrino, Brindisi
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - Unità di Onco-Ematologia - Azienda Ospedaliera - Garibaldi, Catania
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Unità Operativa Oncologia Medica - A.O. Pugliese Ciaccio, Catanzaro
  - Azienda Ospedaliero Universitaria Arcispedale Sant'Anna Dipartimento di Scienze Mediche Sezione di Ematologia e Fisiopatologia dell'Emostasi, Cona
  - U.O. Ematologia - P.O. Annunziata - A.O. di Cosenza, Cosenza
  - Unità di Ricerca e di Malattie del sangue - Ematologia San Luca Vecchio Pad. 16 - 1° Piano, Florence
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Azienda Ospedaliera Universitaria - Policlinico G. Martino Dipartimento di Medicina Interna - U.O. Messina, Messina
  - U.O. Ematologia - P.O. Annunziata - A.O. di Cosenza, Messina
  - UO Ematologia - AOU Policlinico di Modena, Modena
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - U.O. di Oncoematologia -plesso ospedaliero "A. Tortora" di Pagani, Pagani
  - U.O. di Ematologia con trapianto - Centro di Riferimento Regionale per le coagulopatie rare nel bambino e nell'adulto Dipart. Biomedico di Medicina Interna - A.U. Policlinico "Paolo Giaccone", Palermo
  - Day Hospital dell'U.O.C di Ematologia e CTMO Padiglione 1 TORRE DELLE MEDICINE, 6° piano, Parma
  - UOS di Ematologia Servizio di Immunoematologia e medicina Trasfusionale Azienda Sanitaria Provinciale 7, Ragusa
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale "Infermi", Rimini
  - Asl Roma 2, Ospedale S. Eugenio- Ospedale S.Eugenio - Uoc Ematologia, Roma
  - Az. Ospedaliera "Sant' Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Roma
  - Divisione Ematologia - Università Campus Bio-Medico, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - Unità Operativa di Oncologia - Presidio Ospedaliero N. Giannetasio - Azienda ASL 3, Rossano
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ematologia - Dipartimento di Medicina Clinica e Sperimentale, Sassari
  - U.O.C. Ematologia - A.O. Senese - Policlinico " Le Scotte", Siena
  - U.O.C. di Ematolgia - A.O. " SS Annunziata" - P.O. S.G. Moscati, Taranto
  - A.O. Santa Maria - Terni S.C Oncoematologia, Terni
  - Divisione di Ematologia dell' Università degli Studi di Torino - "Città della Salute e della Scienza di Torino", Torino
  - Struttura Complessa II Medicina - Ematologia - Centro di Riferimento Ematologico - Ospedale Maggiore, Trieste
- London North West Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Krepper D, Sparano F, Giesinger JM, Gaidano G, Niscola P, Codeluppi K, Antonioli E, Califano C, Floro L, Annibali O, Fozza C, Tafuri A, Mazza P, Potenza L, Vignetti M, Cavo M, Petrucci MT, Efficace F. Assessing frailty in patients with relapsed/refractory multiple myeloma: A comparison between the patient-reported frailty phenotype and the International Myeloma Working Group frailty index. J Geriatr Oncol. 2025 Jul;16(6):102266. doi: 10.1016/j.jgo.2025.102266. Epub 2025 Jun 4. PMID 40472573
- [Derived] Efficace F, Boccadoro M, Palumbo A, Petrucci MT, Cottone F, Cannella L, Zamagni E, Niscola P, Kyriakou C, Caravita T, Offidani M, Mandelli F, Cavo M. A prospective observational study to assess clinical decision-making, prognosis, quality of life and satisfaction with care in patients with relapsed/refractory multiple myeloma: the CLARITY study protocol. Health Qual Life Outcomes. 2018 Jun 18;16(1):127. doi: 10.1186/s12955-018-0953-4. PMID 29914509